CLINICAL TRIAL: NCT03026127
Title: A Novel Cognitive Reappraisal Intervention for Suicide Prevention
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Stanford University (Other); Florida State University (Other); National Institute of Mental Health (NIMH) (NIH); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1603017115; 5R33MH110542 (NIH); 1R61MH110542 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2017-01-20 (Estimated); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Suicide Prevention
Keywords: Suicide; Middle-aged and Older Adults; Cognitive Reappraisal; Emotion Regulation
MeSH Terms: conditions — Suicide Prevention; Suicide; Emotional Regulation | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRISP (R33) (Experimental): Cognitive Reappraisal Intervention for Suicide Prevention (CRISP) is a psychosocial intervention aimed to reduce suicide risk in middle-aged and older adults who have been hospitalized for suicidal ideation or suicide attempt. CRISP offers a combination of emotion regulation techniques, including changing the subject's perspective or the way he/she thinks to improve emotion reactions. Additional strategies taught include the provision of environmental adaptation tools (notes, checklists, calendars, etc), phone calls, and a tablet application called WellPATH.
  Interventions: Behavioral: Cognitive Reappraisal Intervention for Suicide Prevention
- Supportive Therapy (ST) (R33) (Active Comparator): Supportive Therapy focuses on: 1. facilitating expression of affect; 2. conveying to the patient that he or she is understood; 3. offering empathy; and 4. highlighting positive experiences. The ST manual aims to standardize nonspecific therapeutic factors.
  Interventions: Behavioral: Supportive Therapy
- CRISP (R61) (Experimental): Cognitive Reappraisal Intervention for Suicide Prevention (CRISP) is a psychosocial intervention aimed to reduce suicide risk in middle-aged and older adults who have been hospitalized for suicidal ideation or suicide attempt. CRISP offers a combination of emotion regulation techniques, including changing the subject's perspective or the way he/she thinks to improve emotion reactions. Additional strategies taught include the provision of environmental adaptation tools (notes, checklists, calendars, etc), phone calls, and a tablet application called WellPATH.
  Interventions: Behavioral: Cognitive Reappraisal Intervention for Suicide Prevention

INTERVENTIONS:
Behavioral: Cognitive Reappraisal Intervention for Suicide Prevention — Cognitive Reappraisal Intervention for Suicide Prevention, or CRISP, is a psychosocial intervention aimed to reduce suicide risk in middle-aged and older adults who have been hospitalized for suicidal ideation or suicide attempt. CRISP offers a combination of emotion regulation techniques, including changing the subject's perspective or the way he/she thinks to improve emotion reactions. Additional strategies taught include the provision of environmental adaptation tools (notes, checklists, calendars, etc), phone calls, and a tablet application called WellPATH.
  Other Names: CRISP
  Arms: CRISP (R33); CRISP (R61)
Behavioral: Supportive Therapy — ST focuses on: 1. facilitating expression of affect; 2. conveying to the patient that he or she is understood; 3. offering empathy; and 4. highlighting positive experiences. The ST manual aims to standardize nonspecific therapeutic factors
  Other Names: ST
  Arms: Supportive Therapy (ST) (R33)

SUMMARY:
The goal of this trial is to refine and test a novel emotion-regulation based psychosocial intervention designed to reduce suicide risk in middle-aged and older adults (50-90 years old) who have been discharged after a suicide-related hospitalization (i.e. for suicidal ideation or suicide attempt).

DETAILED DESCRIPTION:
The Investigators developed a novel psychosocial intervention called "Cognitive Reappraisal Intervention for Suicide Prevention (CRISP)," which aims to improve cognitive reappraisal ability (i.e. the ability to modify the appraisal of a situation to alter its emotional significance) (target), and reduce suicide risk (outcome). The conceptual framework views suicidal ideation and behavior as failed attempts to regulate negative emotions and by improving cognitive reappraisal, an effective emotion regulation strategy, the investigators expect to reduce suicide risk. This theory is supported by studies showing that unsuccessful attempts to regulate negative emotions and decreased cognitive reappraisal are associated with increased suicidal ideation and behavior.

The R61 phase is a proof-of-principle phase and its goals are to optimize CRISP and test its engagement with cognitive reappraisal. Certified social workers will administer 12 weekly sessions of CRISP to 40 middle-aged and older adults (50-90 years old) after a suicide-related hospitalization. Research assistants, unaware of the study aims, will conduct assessments at study entry (hospital admission), discharge, 6 and 12 weeks post-discharge. Target engagement will be assessed with EEG assessments during a standard pictured-based stimuli and our novel cognitive reappraisal paradigm.

The R33 phase aims to provide further evidence of target engagement of the optimized CRISP in a larger sample, evaluate the relationship of cognitive reappraisal with suicide risk as measured with Columbia Suicide Severity Rating Scale (C-SSRS) and estimate implementation parameters for a large-scale clinical trial. A different sample of 90 middle-aged and older adults (using the same inclusion/exclusion criteria as for the R61 phase) will be randomized to CRISP or to Supportive Therapy (ST, a control treatment not designed to improve emotion regulation). Assessments will be conducted on admission, at discharge, and at 6, 12 and 24 weeks post-discharge. Primary aims are: 1) CRISP participants will show improvement in cognitive reappraisal ability from discharge to end of treatment; and 2) improvement in cognitive reappraisal ability will be associated with suicide risk over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older
* Diagnosis (based on SCID-5 Clinical Trials Version to assess DSM-5 diagnoses): Any DSM-5 depression or anxiety diagnosis, including major depressive disorder, bipolar depression, depressive disorder Not Elsewhere Classified, anxiety disorder Not Elsewhere Classified, adjustment disorder with anxiety and depressed mood (but without any of the diagnoses shown under Exclusion Criteria)
* Recent hospitalization for suicidal ideation or suicide attempt. At hospital admission, Columbia Suicide Severity Rating Scale greater or equal to 3, "Active Suicidal Ideation with any methods or a suicide attempt."
* Patients with any degree of suicidal ideation at discharge (Columbia Suicide Severity Rating greater or equal to 0) will be included.
* Patients who are on psychotropics and on after-care community psychotherapy will also be included.

Exclusion Criteria:

* History or current diagnosis of Psychotic Disorders; Current Diagnosis of Bipolar I or Bipolar II, with current episode hypomanic, manic or mixed; Diagnosis of Dementia.
* Cognitive Impairment: Mini Mental State Exam (MMSE) < 24.
* Acute or severe medical illness (i.e. delirium; decompensated cardiac, liver, or kidney failure; major surgery; stroke or myocardial infarction during the three months prior to entry.
* Aphasia, sensory problems, and/or inability to speak English.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Institute of Geriatric Psychiatry, Weill Cornell Medicine, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: https://nda.nih.gov/

REFERENCES:
- [Derived] Kiosses DN, Alexopoulos GS, Hajcak G, Apfeldorf W, Duberstein PR, Putrino D, Gross JJ. Cognitive Reappraisal Intervention for Suicide Prevention (CRISP) for Middle-Aged and Older Adults Hospitalized for Suicidality. Am J Geriatr Psychiatry. 2018 Apr;26(4):494-503. doi: 10.1016/j.jagp.2017.11.009. Epub 2017 Dec 27. PMID 29395858

RESULTS

PARTICIPANT FLOW:
Groups:
- CRISP (R61): Experimental: CRISP (R61) Cognitive Reappraisal Intervention for Suicide Prevention (CRISP) is a psychosocial intervention aimed to reduce suicide risk in middle-aged and older adults who have been hospitalized for suicidal ideation or suicide attempt. CRISP offers a combination of emotion regulation techniques, including changing the subject's perspective or the way he/she thinks to improve emotion reactions. Additional strategies taught include the provision of environmental adaptation tools (notes, checklists, calendars, etc), phone calls, and a tablet application called WellPATH.
- CRISP (R33): Experimental: CRISP (R33) Cognitive Reappraisal Intervention for Suicide Prevention (CRISP) is a psychosocial intervention aimed to reduce suicide risk in middle-aged and older adults who have been hospitalized for suicidal ideation or suicide attempt. CRISP offers a combination of emotion regulation techniques, including changing the subject's perspective or the way he/she thinks to improve emotion reactions. Additional strategies taught include the provision of environmental adaptation tools (notes, checklists, calendars, etc), phone calls, and a tablet application called WellPATH.
- CRISP (ST) (R33): Active Comparator: Supportive Therapy (ST) (R33) Supportive Therapy focuses on: 1. facilitating expression of affect; 2. conveying to the patient that he or she is understood; 3. offering empathy; and 4. highlighting positive experiences. The ST manual aims to standardize nonspecific therapeutic factors.
Period: CRISP R61
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33)
Started | 35 | 0 | 0
Completed | 23 | 0 | 0
Not Completed | 12 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Dropped before therapy | 5 | 0 | 0
Period: CRISP R33
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33)
Started | 0 | 48 | 24
Completed | 0 | 17 | 10
Not Completed | 0 | 31 | 14
Not completed — Lost to Follow-up | 0 | 5 | 4
Not completed — Adverse Event | 0 | 9 | 5
Not completed — Withdrawal by Subject | 0 | 9 | 1
Not completed — Lack of Efficacy | 0 | 3 | 2
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Transportation | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33) | Total
Number analyzed (Participants) | 35 | 48 | 24 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.80 (8.47) | 60.94 (8.30) | 60.63 (9.05) | 60.82 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 14 | 66
  Male | 9 | 22 | 10 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 5 | 13
  Not Hispanic or Latino | 29 | 46 | 19 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 5 | 4 | 13
  White | 27 | 40 | 17 | 84
  More than one race | 0 | 3 | 3 | 6
  Unknown or Not Reported | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Late Positive Potential, as Measured by the Electroencephalagram (EEG), Autobiographical Affective Regulation Task (AART), and a Standard Picture-based Emotion Regulation Task. (Only for the R33)
Description: The reported values for each assessment represent μVoltage (a unit of electrical potential) during EEG tasks. These values are the mean result of a composite measure (50% of each task) of μVoltage during the Autobiographical Affective Regulation Task (AART) and a standard picture-based emotion regulation task. Higher values reflect stronger emotional response and lower cognitive reappraisal ability. The results are interpreted comparatively to other values (other groups or other time points) (Only for the R33).
Time Frame: Baseline, 6, 12
Population: This is the analyses of the R33 phase of the study.
Measure: Mean (Standard Deviation); unit: μVoltage
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33)
Number analyzed (Participants) | 0 | 48 | 24
μVoltage
  Baseline: number analyzed (Participants) | 0 | 23 | 14
  Baseline |  | 5.61 (15.97) | 4.38 (9.20)
  Week 6: number analyzed (Participants) | 0 | 13 | 10
  Week 6 |  | 1.51 (9.10) | 0.48 (12.20)
  Week 12: number analyzed (Participants) | 0 | 12 | 6
  Week 12 |  | 2.09 (6.20) | 0.78 (5.22)

2. Primary Outcome: Changes in Electrocortical Measures (i.e., Late Positive Potential, LPP) (Only for the R61)
Description: The reported values for each assessment represent μVoltage (a unit of electrical potential) during EEG tasks at Baseline and Week 12. These values are the mean result of a composite measure (50% of each task) of a) a standardized picture-based emotion regulation task in parietal (Pz) site during 1600-2000ms and b) AART in parietal (Pz) site during 0-3000 ms. Higher values reflect stronger emotional response and lower cognitive reappraisal ability. The results are interpreted comparatively to other values (other groups or other time points) (Only for the R61).
Time Frame: Baseline - Week 12
Population: Analyzed subjects for CRISP R61. Out of 35 participants, 12 participants' data were not used for this analysis: 5 dropped before starting therapy, 5 had adverse event, and 2 were lost to follow up.
Measure: Mean (Standard Deviation); unit: μVoltage
Arm/Group | CRISP (R61) | CRISP (R33) | Supportive Therapy (ST) (R33)
Number analyzed (Participants) | 23 | 0 | 0
μVoltage
  Baseline | 4.99 (4.45) |  |
  Week 12: number analyzed (Participants) | 14 | 0 | 0
  Week 12 | 3.10 (3.33) |  |

3. Other Pre Specified Outcome: Change in Suicide Severity, as Measured by the Columbia Suicide Severity Rating Scale (CSSR-S) (Only for the R33)
Description: The CSSR-S assesses risk for suicide, specifically severity of thoughts, intensity of thoughts, behavior and lethality. Questions are scored in categories, 1-5, with lower numbers indicating less severity and higher numbers more severity.
  The outcome variable is scored with respect to the most severe type of ideation from the following Yes or No questions "Wish to be Dead," "Non-Specific Active Suicidal Thoughts," "Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act," "Active Suicidal Ideation with Some Intent to Act, without Specific Plan," and "Active Suicidal Ideation with Specific Plan and Intent." A response of "Yes" yields a score of 1 and a response of "No" yields a score of 0.
  The highest score a participant can receive is 5.
  If the answer to question 2 is "Yes" then questions 3, 4, and 5 are asked. Only if the questions 1 and 2 are recorded as "Yes' the outcome the Intensity of Ideation is completed.
Time Frame: Baseline - Week 12
Population: This analysis is for R33 participants only. R33 participants who did not complete Week 12 were excluded from analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33)
Number analyzed (Participants) | 0 | 19 | 12
score on a scale |  | 0.21 (0.98) | -0.500 (1.45)

ADVERSE EVENTS:
Time Frame: CRISP R61 (12 Weeks) CRISP R33 (24 Weeks)
Arm/Group | CRISP (R61) | CRISP (R33) | CRISP (ST) (R33)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/48 | 0/24
Serious Adverse Events (participants affected / at risk) | 8/35 | 13/48 | 4/24
Other Adverse Events (participants affected / at risk) | 0/35 | 2/48 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRISP (R61) (N=35) | CRISP (R33) (N=48) | CRISP (ST) (R33) (N=24)
Major Depressive Disorder (Psychiatric disorders) | 4 (4) | 9 (10) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRISP (R61) (N=35) | CRISP (R33) (N=48) | CRISP (ST) (R33) (N=24)
Psychiatric Episode (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol: Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03026127/Prot_000.pdf
  • Study Protocol: Intervention Manual (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03026127/Prot_001.pdf
  • Informed Consent Form: CRISP R33 ICF (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03026127/ICF_002.pdf
  • Informed Consent Form: CRISP R61 ICF (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03026127/ICF_003.pdf